CLINICAL TRIAL: NCT04937426
Title: Development of a Laboratory Test for the Detection of a Fluorescent-labeled Urease Inhibitor Marker Attached to Helicobacter Pylori Using Biopsies Taken During Gastroscopy in Patients in Which the Bacterium is Suspected
Brief Title: Development of a Laboratory Test for the Detection of a Fluorescent-labeled Urease Inhibitor Marker Attached to Helicobacter Pylori
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0085-20
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Helicobacter Pylori

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescent-labeled Urease Inhibitor Marker to Detect Helicobacter Pylori (Experimental): During gastroscopy additional biopsies are taken in cases where infection with helicobacter pylori is suspected. It will then undergo laboratory analysis with fluorescent-labeled urease inhibitor marker. Results will be compared to standard analysis to determine efficacy.
  Interventions: Diagnostic Test: Fluorescent-labeled Urease Inhibitor Marker to Detect Helicobacter Pylori

INTERVENTIONS:
Diagnostic Test: Fluorescent-labeled Urease Inhibitor Marker to Detect Helicobacter Pylori — Diagnostic laboratory test for detection of helicobacter pylori

SUMMARY:
The aim of this study is to compare the usual rapid urease test (RUT) to a new florescent-labeled urease inhibitor marker to diagnose Helicobacter Pylori.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastroendoscopy with suspected Helicobacter Pylori

Exclusion Criteria:

* Patients with active bleeding
* Patients treated with anti-coagulation medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a Fluorescent-labeled Urease Inhibitor Marker to Detect Helicobacter Pylori Infection | Two years
  Comparison of results of biopsies analyzed with a fluorescent-labeled urease inhibitor marker to detect Helicobacter Pylori infection and results will be compared to standard tests to detect Helicobacter Pylori

CONTACTS AND LOCATIONS:
Overall Officials: Yael Kopelman, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No